CLINICAL TRIAL: NCT03694288
Title: The FIRM Trial - A Randomized Clinical Trial Evaluating Fixation In-situ vs Removal for Midfoot Lisfranc Injuries
Brief Title: Fixation In-situ vs Removal for Midfoot Lisfranc Injuries
Acronym: FIRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Prism Schneider, Orthopaedic Trauma Research Lead, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIRM Protocol
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Lisfranc Injuries
Keywords: Lisfranc
MeSH Terms: interventions — Device Removal

STUDY DESIGN:
Intervention Model Description: This study is a multicenter randomized clinical trial comparing implant retention (Retention) to scheduled removal of implants (Removal) in skeletally mature patients with previously operatively treated Lisfranc injuries requiring screw and/or plate fixation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removal Group (Active Comparator): The implant removal group will have surgery scheduled 6 months after their initial surgical fixation.
  Interventions: Procedure: Implant removal
- Retention Group (No Intervention): The implant retention group will retain their implant for a minimum of 2 years from the time of their initial surgery.

INTERVENTIONS:
Procedure: Implant removal — Surgical Implant removal
  Arms: Removal Group

SUMMARY:
Injuries to the midfoot tarsometatarsal joint, or Lisfranc joint, are notoriously debilitating. Poor functional outcomes following Lisfranc injuries have motivated surgeons to look for potential improvements in post-operative care. There are currently no evidence-based guidelines to direct implant removal for patients with operatively treated Lisfranc injuries. Routine implant removal has significant implications related to health care costs, lost time from work, potential surgical complications, and possibly functional impairment. Therefore, stakeholders including patients, surgeons, employers, and administrators will benefit from evidence-based guidelines for implant removal following operatively treated Lisfranc injuries. To date, there has not been a prospective randomized study evaluating the efficacy of implant removal compared with implant retention for Lisfranc injuries. The aim of this study is to directly compare patient-reported and radiographic outcomes, in order to provide robust evidence for optimal post-operative treatment regimens regarding implant removal or retention for operatively treated Lisfranc injuries.

DETAILED DESCRIPTION:
This study is a multicenter, randomized clinical trial comparing implant retention (Retention Group) to scheduled implant removal (Removal Group) in 100 skeletally mature patients with Lisfranc injuries previously treated with screw and/or plate fixation. The primary outcome measure is the validated, patient-reported Foot and Ankle Ability Measure (FAAM) at 1-year post initial Lisfranc injury. Secondary outcome measures include: 1. American Orthopedics Foot and Ankle Midfoot Score (AOFAS), 2. patient-reported Visual Analogue Scale (VAS) for Foot and Ankle, 3. range of motion, 4. radiographic assessment of Lisfranc reduction, 5. comparative cost analysis between treatment groups. This study will follow patients for 1-year post-injury.

Patients, surgeons, employers, and administrators will benefit from an evidence-based approach to implant removal following operatively treated Lisfranc injuries. This study will allow orthopaedic surgeons to counsel patients regarding the advantages and disadvantages of implant retention compared with removal. This study will provide robust data to inform clinical decision making for surgeons and provide patients with information regarding expected functional outcomes following Lisfranc injuries.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and skeletally mature
* Subject has Lisfranc injury that was previously treated with screws and/or plate fixation within 21 days of initial injury
* Subject must be enrolled in study within 6 weeks (+/-2 weeks) from time of initial fixation operation
* The patient must be medically fit for anaesthesia
* Subject is willing and able to provide written informed consent for trial participation
* Subject is willing and able to comply with the study protocol including return for all follow-up evaluations

Exclusion Criteria:

* Subject has a significant pre-existing foot injury or deformity
* There has been loss of fixation or reduction prior to enrollment
* Subject was treated with a primary tarsometatarsal joint fusion
* Subject has a delay in initial treatment greater than 21 days from time of injury
* Subject has an active infection in the area of surgical approach
* Subject has concomitant injury which, in the opinion of the attending surgeon, is likely to impair rehabilitation or prolong fracture healing time
* Subject has a history of rheumatoid arthritis, Diabetes, metabolic bone disease (including osteoporosis actively being treated), active malignancy, pathologic fracture or other pre-existing pathologic condition affecting the Lisfranc complex
* Subject has a high risk of death from surgery (ASA physical status Class V)
* Subject is likely unable to maintain follow-up
* Subject has cognitive impairment or language difficulties that would impede the valid completion of questionnaires
* Subject is pregnant or planning on becoming pregnant in the following year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | 24 months
  FAAM is a patient-reported outcome tool used to assess physical function at 24 months post initial Lisfranc surgery. This instrument includes 2 sub-scales: activities of daily living sub scale of 21 items and sport sub scale of 8 items. Answers for both scales are based on a Likert scale (4-0) of: 4) No difficulty, 3) Slight difficulty, 2) Moderate difficulty, 1) Extreme difficulty, and 0) Unable to do. Questions for which "N/A" is indicated are not counted. Two scores are reported, one for each sub scale. To calculate the score for either sub scale, the total number of points are added, divided by the number of possible points (84 for ADL and 32 for sports), and multiplied by 100. Higher scores reflect a higher level of physical function.

SECONDARY OUTCOMES:
American Orthopedics Foot and Ankle Midfoot Score (AOFAS) | 24 months
  AOFAS is a surgeon-administered questionnaire, used for assessment of pain, function and alignment. The total score is reported. Scores range from 0 to 100, with a healthy midfoot receiving 100 points
Patient-reported Visual Analogue Scale (VAS) for Foot and Ankle | 24 months
  VAS for Foot and Ankle is a validated tool for assessing pain intensity specific to foot injuries. The patient is asked to mark their current situation on a 10 cm line with anchor statements on the left (negative outcome) and on the right (positive outcome). Longer distances (from the "negative outcome" anchor point) represent a better outcome.
Range of motion (ROM) | 24 months
  Assessed buy surgeon
Radiographic assessment of Lisfranc reduction | 24 months
  Maintenance of reduction and degree of arthritic changes across Lisfranc complex (gap between 1st and 2nd metatarsals, between the lateral aspect of the medial cuneiform to the medial aspect of second metatarsal) will be assessed by comparison of index Xrays upon enrollment and follow-up X-rays.
Comparative cost analysis between treatment groups | 24 months
  Comparative cost of treatment and any complications plus incremental costs up to 2-year follow-up will be collected and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada